CLINICAL TRIAL: NCT00136695
Title: Anastrozole Administration in Elderly Hypogonadal Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Benjamin Leder, MD, Principal Invesitgator (MD), Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG0035; 5R01AG025099-05 (NIH); 1R01AG025099-1A1
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Hypogonadism
Keywords: Aging
MeSH Terms: conditions — Hypogonadism | interventions — Anastrozole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- anastrozole (Experimental): anastrozole
  Interventions: Drug: anastrozole
- placebo (Placebo Comparator): placebo
  Interventions: Drug: anastrozole

INTERVENTIONS:
Drug: anastrozole — 1 mg QD
  Other Names: arimidex

SUMMARY:
The purpose of the study is to assess the effects of sustained aromatase inhibitor therapy to reduce estrogen levels in elderly men with mild hypogonadism (a decreased level of sex hormones).

DETAILED DESCRIPTION:
It has long been accepted that aging in men is associated with a slow, steady decline in gonadal androgen (male sex hormone) production. Several studies have explored androgen replacement, but the safety and efficacy of testosterone administration remains controversial. Aromatase inhibitors may provide a particularly useful way to restore normal androgen production in aging men.

This study will recruit 150 male volunteers, 60 years of age or older, to be randomized to receive either anastrozole or a placebo for 24 months. Six visits are planned over the 96-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Men ages 60 and older
* Serum testosterone between 150-300 ng/dL
* Symptoms suggestive of androgen deficiency

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Z. Leder, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- General Clinical Research Center, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Leder BZ, Rohrer JL, Rubin SD, Gallo J, Longcope C. Effects of aromatase inhibition in elderly men with low or borderline-low serum testosterone levels. J Clin Endocrinol Metab. 2004 Mar;89(3):1174-80. doi: 10.1210/jc.2003-031467. PMID 15001605
- [Background] Taxel P, Kennedy DG, Fall PM, Willard AK, Clive JM, Raisz LG. The effect of aromatase inhibition on sex steroids, gonadotropins, and markers of bone turnover in older men. J Clin Endocrinol Metab. 2001 Jun;86(6):2869-74. doi: 10.1210/jcem.86.6.7541. PMID 11397902

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anastrozole | Placebo
Started | 45 | 43
Completed | 34 | 35
Not Completed | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anastrozole | Placebo | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (4) | 66 (4) | 66 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 34 | 35 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change in Lean Body Mass
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 34 | 35
grams | -2000 (1000) | -1500 (500)

ADVERSE EVENTS:
Arm/Group | Anastrozole | Placebo
Serious Adverse Events (participants affected / at risk) | 4/34 | 1/35
Other Adverse Events (participants affected / at risk) | 3/34 | 3/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole (N=34) | Placebo (N=35)
prostate cancer (Renal and urinary disorders) | 0 | 1
pancreatic cancer (Endocrine disorders) | 1 | 0
hepatitis A (Gastrointestinal disorders) | 1 | 0
pulmonary embolism (Blood and lymphatic system disorders) | 1 | 0
embolic stroke (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole (N=34) | Placebo (N=35)
PSA increase (Renal and urinary disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No